CLINICAL TRIAL: NCT04543344
Title: A Phase 1, Randomized, Parallel-Group Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Single or Multiple Subcutaneous Doses of Lyophilized Formulation of Recifercept in Healthy Participants
Brief Title: Study To Evaluate The Pharmacokinetic, Safety And Tolerability Of Single Or Multiple Subcutaneous Doses of Recifercept
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C4181004; 2020-000545-14 (EudraCT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only cohort 1 of the study is blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Repeated multiple doses
  Interventions: Drug: Recifercept
- placebo (Placebo Comparator): Repeated multiple doses
  Interventions: Other: Placebo
- High Dose (Experimental): Repeated multiple doses
  Interventions: Drug: Recifercept

INTERVENTIONS:
Drug: Recifercept — recifercept powder for solution for injection
  Other Names: PF-07256472
  Arms: High Dose; Low Dose
Other: Placebo — solution for injection
  Arms: placebo

SUMMARY:
This will be a single center, randomized, parallel group, repeated dose study of recifercept (Cohort 1 and Cohort 2) or placebo (only in Cohort 1) in approximately 18 healthy participants, using 2 cohorts (N = 9) at two dose levels of recifercept.

ELIGIBILITY:
Inclusion Criteria:

* Male participants and female participants of nonchildbearing potential
* Participants who are overtly healthy
* Capable of giving signed informed consent

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 312 and 504 hours post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | 0, 2, 4, 6, 12, 24, 48 and 72 hours post-dose
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau)
Maximum Observed Plasma Concentration (Cmax) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 312 and 504 hours post-dose
  Maximum Observed Plasma Concentration directly from data
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 312 and 504 hours post-dose
  Time to reach Cmax
Plasma Decay Half-Life (t1/2) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 312 and 504 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Accumulation Ratio (Rac) | 0, 2, 4, 6, 12, 24, 48 and 72 hours post-dose
  Accumulation ratio was calculated as, Rac obtained from Area Under the Concentration Time Curve (AUC) from time 0-t (Day X) divided by AUC from time 0-t (Day 1).

SECONDARY OUTCOMES:
Incidence of Anti-drug antibodies (ADA) | 6 months post-dose
  Incidence of participants who are ADA positive
Incidence of Neutralizing antibodies (NAb) | 6 months post-dose
  Incidence of participants who are NAb positive

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4181004